CLINICAL TRIAL: NCT06680583
Title: Utilizing of Physiological Parameters And Derived Indices to Predict The Prognosis of Cirrhotic Patients With Gastrointestinal Bleeding
Brief Title: Utilizing of Physiological Parameters Predict the Prognosis of Cirrhotic Patients With Gastrointestinal Bleeding
Acronym: SI
Status: Recruiting | Type: Observational
Sponsor: St. Martin De Porress Hospital (Other)
Responsible Party: Principal Investigator, Chia-hsi Chen, Emergency and Critical Care Physician, St. Martin De Porress Hospital
Other Study IDs: St. Martin De Porres Hospital; physical parameters (Registry Identifier: physical parameters)
Record Dates: First submitted 2024-11-04; First posted 2024-11-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Liver Cirrhosis; Gastrointestinal Bleeding
Keywords: cirrhosis; gastrointestinal bleeding; physical indicator; shock index
MeSH Terms: conditions — Liver Cirrhosis; Gastrointestinal Hemorrhage; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cirrhosis: cirrhosis with gastrointestinal bleeding
  Interventions: Other: physical indicators such as shock index relatives

INTERVENTIONS:
Other: physical indicators such as shock index relatives — shock index relatives indicators used in the prediction of cirrhosis with gastrointestinal bleeding
  Other Names: MSI, Age SI, RASI

SUMMARY:
Can physiological indicators such as quick Sequential Organ Failure Assessment , Shock Index, and its derived indicators such as Modified Shock Index , Age Shock Index and Respiratory Adjusted Shock Index accurately predict the prognosis of cirrhosis patients with gastrointestinal bleeding? To explore the improvement of emergency and critical care patient management.

DETAILED DESCRIPTION:
Cirrhosis is a common chronic liver disease with gastrointestinal bleeding being one of its complications. Gastrointestinal bleeding is quite common in patients with cirrhosis, but its prognosis is difficult to accurately predict. In current clinical practice, critical care physicians often use physiological indicators to assess the risk level of patients. Among them, the Shock Index and its derived indicators such as the Modified Shock Index, Age Shock Index, and Respiratory Adjusted Shock Index have been widely used in other fields, but their actual value in patients with cirrhosis complicated by gastrointestinal bleeding is not yet clear.

The prognosis of cirrhosis patients with gastrointestinal bleeding affects the quality of life and survival of the patients, thus necessitating the establishment of a reliable prognostic assessment tool to assist critical care physicians in making rapid treatment decisions. The motivation of this study is to explore the application value of Shock Index-related indicators in predicting the prognosis of cirrhosis patients with gastrointestinal bleeding, in order to improve the medical efficiency for this specific group of critically ill patients.

ELIGIBILITY:
Inclusion Criteria: cirrhosis with gastrointestinal bleeding -

Exclusion Criteria: no complete medical record and trauma patient

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cirrhosis with gastrointestinal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
shock index= heart rate / systolic blood pressure normal range:0.5-0.7 Modified shock index = heart rate/mean arterial pressure(MAP) age shock index = SI x age number respiratory adjusted shock index(RASI) = HR/SBP × RR/10. MAP = DP + 1/3(SP - DP) | through study completion, an average of 6 months
  find the shock index relatives indicators in the prognosis prediction of cirrhosis with gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Chin Jou Jou, professor, Study Director — St. Martin De Porres Hospital Education and Research
Locations (1):
- St. Martin De Porres Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
This study include the medical privacy of cirrhosis.

REFERENCES:
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/34812069/ — Physical indicators with shock index relatives are used in the prediction of prognosis on cirrhosis with gastrointestinal bleeding